CLINICAL TRIAL: NCT04516733
Title: Precoce Medical Care by the Mobil Support for Patients With Glioblastoma Receiving Specific Medical Oncology Treatment
Brief Title: Precoce Medical Care by the Mobil Support for Patients With Glioblastoma
Acronym: GLIOSUPPORT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut du Cancer de Montpellier - Val d'Aurelle (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: PROICM 2018-04 GLI
Record Dates: First submitted 2020-08-11; First posted 2020-08-18 (Actual); Last update posted 2022-03-14 (Actual); Status verified 2022-03

CONDITIONS: Glioblastoma
Keywords: supportive care; mobil unit
MeSH Terms: conditions — Glioblastoma | interventions — Palliative Care

STUDY DESIGN:
Intervention Model Description: in addition to oncology care, there will be a care with palliative team and neuropsychological care
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- single arm (Other): patient with glioblastoma
  Interventions: Other: supportive care

INTERVENTIONS:
Other: supportive care — visit with supportiv unit and neuropsychologue every 3 months

SUMMARY:
Most patients with glioblastoma have impaired cognitive function, autonomy, and quality of life.

This clinical situation, combined with a limited life expectancy, makes the preservation of quality of life a major objective, in a supportive environment that respects family integration. This is especially true since there is an established relationship between health-related quality of life, as measured by questionnaires.

In this context, and despite the lack of impact on overall survival, improving quality of life becomes a priority objective in recent Phase III trials.

The feasibility of introducing early accompaniment in GBM should be assessed in the diagnostic and therapeutic announcement environment. In order to measure the expected impact as favorable in the patient and his family, a broad survey of the classic domains of quality of life and more specifically dedicated to neurological symptomatology.

DETAILED DESCRIPTION:
glioblastomas are the most common primary malignant tumours of the central nervous system.They represent about 2000 new cases per year in France.

Despite active treatments including surgery, radiotherapy and chemotherapy, patient survival is limited without possible cure.

Most patients with glioblastoma have impaired cognitive function, autonomy, and quality of life. Exploration of verbal memory in these patients shows that its deterioration is correlated with a more unfavourable prognosis, after adjustment with other usual prognostic factors.

This clinical situation, combined with a limited life expectancy, makes the preservation of quality of life a major objective, in a supportive environment that respects family integration. This is especially true since there is an established relationship between health-related quality of life, as measured by questionnaires.

The feasibility of introducing early accompaniment in GBM should be assessed in the diagnostic and therapeutic announcement environment. In order to measure the expected impact as favorable in the patient and his family, a broad survey of the classic domains of quality of life and more specifically dedicated to neurological symptomatology.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient ( ≥ 18 years),
* Histological diagnosis of Glioblastoma
* Oncology caret at ICM (regardless of treatment: Stupp protocol, chemotherapy alone, targeted therapy, etc.);
* Patient consent signed after informed information.

Exclusion Criteria:

* Patient unable to consent to the study
* Major impairment of the general health : performance status OMS =4;
* Patient not affiliated with a French social security

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2019-05-10 (Actual); Primary Completion 2020-09-15 (Actual); Study Completion 2022-02-15 (Actual)

PRIMARY OUTCOMES:
Assess the feasibility in terms of compliance with early medical care in glioblastoma patients by palliative care unit. | from date of inclusion visit until an average of 3 months
  Compliance is defined as the proportion of patients attending three palliative care unit visits (Ve1, Ve2 and Ve3).

SECONDARY OUTCOMES:
The recruitment rate (proportion of patients giving consent to participate in the study among eligible patients during screening) | at the inclusion visit
  Participation rate, defined as the proportion of patients who accepted inclusion in the study among all screened patients. Investigator expect an 80% participation rate in this study
Proportion of patients completing all quality of life assessments (QLQ-C30 (Quality Life Questionnaire) at palliative care unit visits (Ve1, Ve2 and Ve3) | from date of inclusion visit until an average of 3 months
  The proportion of palliative care unit consultations not carried out due to impossibility for the palliative care unit
Proportion of patients completing all BN20 assessments (Brain Cancer Module) at palliative care unit visits (Ve1, Ve2 and Ve3) | from date of inclusion visit until an average of 3 months
  The proportion of palliative care unit consultations not carried out due to impossibility for the palliative care unit
Proportion of patients completing all anxiety assessments (HADS, Hospital Anxiety and Depression Scale) at palliative care unit visits (Ve1, Ve2 and Ve3) | from date of inclusion visit until an average of 3 months
  The proportion of palliative care unit consultations not carried out due to impossibility for the palliative care unit
Changes over time in patients' quality of life | from date of inclusion visit until an average of 3 months
  Score of questionnaire (QLQ-C30 (Quality Life Questionnaire)
Changes over time in patients' quality of life | from date of inclusion visit until an average of 3 months
  Score of questionnaire BN20 (Brain Cancer Module)
The evolution over time of anxiety and depressive affects in patients | from date of inclusion visit until an average of 3 months
  score of HADS questionnaire (Hospital Anxiety and Depression Scale). <9 no significant, between 10 and12 limit and > 13 significant
The evolution over time of neurocognitive performance in patients and the delay before neurocognitive degradation (Mattis DRS scale); | from date of inclusion visit until an average of 3 months
  Neurocognitive performance of patients assessed by total score and scores at sub-scales of attention, initiation, conceptualization, construction and memory at the Mattis DRS scale
Rate of patients who have written advance directives since the diagnostic announcement; | From date of inclusion until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 100 months
  The percentage of patients for whom advance directives have been written and documented in the medical record,
Rate of patients who have designated a support person since the diagnostic announcement | From date of inclusion until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 100 months
  the percentage of patients for whom the support person has been designated
proportion of patients receiving specific medical oncology treatment in their last month of life | From date of inclusion until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 100 months
  Percentage of patients receiving specific oncology treatment in the month prior to death
Overall survival | From date of inclusion until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 100 months
  defined as the delay between the date of inclusion and the date of death (any cause) or the date of last update
The proportion of patients diagnosed with glioblastoma that are available for this medical care | at the inclusion visit
  Percentage of patients diagnosed with glioblastoma not care at the center during the inclusion period will be reported, as well as the reasons for not cared at the ICM center

CONTACTS AND LOCATIONS:
Overall Officials: Michel FABBRO, MD, Study Chair — Institut du Cancer de Montpellier - Val d'Aurelle
Locations (1):
- ICM Val d'Aurelle, Montpellier, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Aaronson NK, Ahmedzai S, Bergman B, Bullinger M, Cull A, Duez NJ, Filiberti A, Flechtner H, Fleishman SB, de Haes JC, et al. The European Organization for Research and Treatment of Cancer QLQ-C30: a quality-of-life instrument for use in international clinical trials in oncology. J Natl Cancer Inst. 1993 Mar 3;85(5):365-76. doi: 10.1093/jnci/85.5.365. PMID 8433390
- [Result] Batchelor TT, Mulholland P, Neyns B, Nabors LB, Campone M, Wick A, Mason W, Mikkelsen T, Phuphanich S, Ashby LS, Degroot J, Gattamaneni R, Cher L, Rosenthal M, Payer F, Jurgensmeier JM, Jain RK, Sorensen AG, Xu J, Liu Q, van den Bent M. Phase III randomized trial comparing the efficacy of cediranib as monotherapy, and in combination with lomustine, versus lomustine alone in patients with recurrent glioblastoma. J Clin Oncol. 2013 Sep 10;31(26):3212-8. doi: 10.1200/JCO.2012.47.2464. Epub 2013 Aug 12. PMID 23940216
- [Result] Brown PD, Ballman KV, Rummans TA, Maurer MJ, Sloan JA, Boeve BF, Gupta L, Tang-Wai DF, Arusell RM, Clark MM, Buckner JC. Prospective study of quality of life in adults with newly diagnosed high-grade gliomas. J Neurooncol. 2006 Feb;76(3):283-91. doi: 10.1007/s11060-005-7020-9. PMID 16163448
- [Result] Cella DF, Tulsky DS, Gray G, Sarafian B, Linn E, Bonomi A, Silberman M, Yellen SB, Winicour P, Brannon J, et al. The Functional Assessment of Cancer Therapy scale: development and validation of the general measure. J Clin Oncol. 1993 Mar;11(3):570-9. doi: 10.1200/JCO.1993.11.3.570. PMID 8445433
- [Result] Chinot OL, Wick W, Mason W, Henriksson R, Saran F, Nishikawa R, Carpentier AF, Hoang-Xuan K, Kavan P, Cernea D, Brandes AA, Hilton M, Abrey L, Cloughesy T. Bevacizumab plus radiotherapy-temozolomide for newly diagnosed glioblastoma. N Engl J Med. 2014 Feb 20;370(8):709-22. doi: 10.1056/NEJMoa1308345. PMID 24552318
- [Result] Darlix A, Zouaoui S, Rigau V, Bessaoud F, Figarella-Branger D, Mathieu-Daude H, Tretarre B, Bauchet F, Duffau H, Taillandier L, Bauchet L. Epidemiology for primary brain tumors: a nationwide population-based study. J Neurooncol. 2017 Feb;131(3):525-546. doi: 10.1007/s11060-016-2318-3. Epub 2016 Nov 16. PMID 27853959
- [Result] Flechl B, Ackerl M, Sax C, Dieckmann K, Crevenna R, Gaiger A, Widhalm G, Preusser M, Marosi C. Neurocognitive and sociodemographic functioning of glioblastoma long-term survivors. J Neurooncol. 2012 Sep;109(2):331-9. doi: 10.1007/s11060-012-0897-1. Epub 2012 May 29. PMID 22644537
- [Result] Flechl B, Sax C, Ackerl M, Crevenna R, Woehrer A, Hainfellner J, Preusser M, Widhalm G, Kiesel B, Lutgendorf-Caucig C, Dieckmann K, Steffal C, Marosi C, Hassler MR. The course of quality of life and neurocognition in newly diagnosed patients with glioblastoma. Radiother Oncol. 2017 Nov;125(2):228-233. doi: 10.1016/j.radonc.2017.07.027. Epub 2017 Aug 8. PMID 28801008
- [Result] Gilbert MR. Antiangiogenic Therapy for Glioblastoma: Complex Biology and Complicated Results. J Clin Oncol. 2016 May 10;34(14):1567-9. doi: 10.1200/JCO.2016.66.5364. Epub 2016 Mar 21. No abstract available. PMID 27001588
- [Result] Gilbert MR, Dignam JJ, Armstrong TS, Wefel JS, Blumenthal DT, Vogelbaum MA, Colman H, Chakravarti A, Pugh S, Won M, Jeraj R, Brown PD, Jaeckle KA, Schiff D, Stieber VW, Brachman DG, Werner-Wasik M, Tremont-Lukats IW, Sulman EP, Aldape KD, Curran WJ Jr, Mehta MP. A randomized trial of bevacizumab for newly diagnosed glioblastoma. N Engl J Med. 2014 Feb 20;370(8):699-708. doi: 10.1056/NEJMoa1308573. PMID 24552317